CLINICAL TRIAL: NCT07094854
Title: Clinical Performance and Antibacterial Effect of a Bulk Fill Alkasite Bioactive Material in Restoring Pulpotomized Primary Molars(Randomized Controlled Clinical Trial)
Brief Title: Clinical Performance and Antibacterial Effect of Alkasite Bioactive Material in Restoring Pulpotomized Primary Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Noha Fouad (Other)
Responsible Party: Sponsor-Investigator, Noha Fouad, Assistant lecturer of Pediatric Dentistry, Faculty of Dentistry, Alexandria University, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Noha Fouad
Record Dates: First submitted 2025-06-29; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Healthy Children
Keywords: Cention Forte; Alkasite; bioactive; pulpotomy; primary teeth; stainless steel crown; bulk fill

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor, statistician and the microbiologist are blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cention forte material (Experimental)
  Interventions: Other: Cention Forte alkasite bioactive restorative material
- Stainless steel crown (Active Comparator)
  Interventions: Other: Stainless steel crown

INTERVENTIONS:
Other: Cention Forte alkasite bioactive restorative material — Cention forte material will be used as a final restoration for pulpotomized second primary molars
  Arms: Cention forte material
Other: Stainless steel crown — The control group using the gold standard stainless steel crown (SSC) as a final restoration for pulpotomized second primary molars
  Arms: Stainless steel crown

SUMMARY:
The study aims to evaluate the clinical performance of Cention-Forte (CF) material in the restoration of pulpotomized second primary molars compared to conventional stainless steel crowns (SSC), and also to assess the restorations' antibacterial effect on salivary cariogenic bacterial count.

DETAILED DESCRIPTION:
A two-arm randomized controlled clinical trial. A total of 40 healthy cooperative children aged 5-9 years, will be selected from the Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Alexandria University, Egypt. Each child selected will have second primary molar with occluso-proximal carious lesions indicated for pulpotomy. Written informed consent will be obtained from their guardians. After the MTA pulpotomy procedure, participants will be randomly allocated into two groups according to the restoration used. Group I (test group n=20) will receive Cention Forte material, while group II (control group n=20) will receive conventional SSC. Using Modified Ryge's Criteria, the clinical performance of the restorations will be evaluated at 1 week and then after 3, 6 and 12 months for marginal adaptation, proximal contact, retention, gross fracture, occlusal wear, surface roughness and secondary caries. Periapical radiographs will be taken at baseline and after 6 and 12 months. Also, the antibacterial effect of the restorations on salivary cariogenic bacterial count will be assessed at baseline and after 1 week, 1 month and 3 months. Plaque and Gingival index scores as well as parental and child's satisfaction will be recorded.

Data will be collected, tabulated, and statistically analysed to obtain the results and conclusions of this study.

ELIGIBILITY:
Inclusion Criteria:

* Cooperative children (Positive or definitely positive) according to the Frankl's behaviour rating scale.
* Children free of any systemic disease or special health care needs (ASA1).
* Completion of an informed consent to participate in the study.
* Second primary molar tooth with occluso-proximal carious lesions indicated for pulpotomy.
* Restorable tooth.
* Radiographically at least two-thirds of the root length is present.
* Presence of neighboring and opposing teeth.

Exclusion Criteria:

* Clinical signs or symptoms of irreversible pulpitis or non- vitality.
* Radiographic signs of degeneration including internal or external root resorption, furcation involvement.
* Pathologic mobility detected by placing the points of a pair of tweezers in the occlusal fossa and gently rocking the tooth buccolingually.
* Reported usage of local or systemic antibiotics, chlorhexidine or fluoride mouthwashes within the last 2 weeks.
* Child with parafunctional habits.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Clinical performance of the restorations using Modified Ryge's Criteria | One year
  The clinical evaluation of the two restorations will be done using parameters of marginal adaptation, proximal contact, retention, gross fracture, occlusal wear, surface roughness, and secondary caries as per the modified United States Public Health Service (USPHS) Ryge's criteria.
  Scores for the modified Ryge's criteria are as follow:
  * alpha: represents the ideal or excellent condition of a restoration
  * bravo: indicates a clinically acceptable restoration with minor defects
  * charlie: indicates restoration is unacceptable clinically and should be replaced
The antibacterial effect of both restorations on salivary cariogenic bacterial count. | 3 months
  The saliva samples will be collected to assess microbiological colony count of S.mutan and lactobacilli at baseline, after 1 week, 1 month and 3 months.

SECONDARY OUTCOMES:
Radiographic success of pulpotomized second primary molars in both groups | One year
  The success of pulpotomy procedure will be assessed radiographically using digital periapical xray after 6 and 12 months.
Gingival index | One year
  Gingival health will be assessed clinically at baseline, then after 3, 6 and 12 months using the gingival index score:
  Scores for the index indicate:
  0: normal gingival
  1. mild inflammation, sllight change in colour and slight edema. No bleeding on probing
  2. Moderate inflammation: redness, edema and glazing. Bleeding on probing.
  3. Severe inflammation: marked redness, edema and ulcerations. Tendency towards spontaneous bleeding
Plaque index | One year
  Gingival health will be assessed clinically using plaque index at baseline, then after 3, 6 and 12 months.
  Plaque index scores indicate:
  0: No plaque
  1. A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in-situ only after application of disclosing solution or by using the probe on the tooth surface
  2. Moderate accumulation of soft deposits within the gingival pocket, or the tooth and gingival margin which can be seen by the naked eye
  3. Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
Child satisfaction | Over one year
  The patient's perception of the treatment will be assessed by using the Facial Image Scale (FIS) that represents satisfaction, indifference, or dissatisfaction. A few minutes will be spent before each procedure to establish rapport with the child and to obtain some notion of the child's understanding of the meaning of those schematic facial expressions. After treatment, the child will be instructed to choose the face that best represented how he/she felt during the procedure.
Parental satisfaction | Over one year
  Parental satisfaction level will be assessed immediately after the procedure with 5-point Likert scale where 1-very dissatisfied; 2-dissatisfied; 3-neutrally satisfied; 4-satisfied; 5-very satisfied. Parents will be asked to rate their satisfaction regarding appearance, color, size, durability, and overall satisfaction for the restoration/crown.

CONTACTS AND LOCATIONS:
Overall Officials: Magda M ElTekeya, Study Director — Alexandria University; Niveen S Bakry, Study Director — Alexandria University; Azza Zakaria, Study Director — Alexandria University
Locations (2):
- Egypt (2):
  - Faculty of Dentistry, Alexandria University, Alexandria
  - Faculty of Pharmacy, Alexandria University, Alexandria

IPD SHARING:
Plan to Share IPD: No